CLINICAL TRIAL: NCT03977480
Title: A Multicenter, Randomized, Double-blind, Placebo Parallel Controlled Clinical Study on the Effecacy and Safety of Different Dosing Regimens of Hemay007 in Patients With Active Ulcerative Colitis
Brief Title: Phase II Study of Hemay007 in Patients With Active Ulcerative Colitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to the difficulty to recruit enough patients, the study was terminated.
Sponsor: Tianjin Hemay Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Ganzhou Hemay Pharmaceutical Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HM007UC2S01
Record Dates: First submitted 2019-04-27; First posted 2019-06-06 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Hemay007 400 mg BID group (Active Comparator): Patients will orally take Hemay007 tablets 400 mg BID for 12 weeks.
  Interventions: Drug: Hemay007
- Hemay007 800 mg QD group (Active Comparator): Patients will orally take Hemay007 tablets 800 mg QD for 12 weeks.
  Interventions: Drug: Hemay007
- Hemay007 600 mg BID group (Active Comparator): Patients will orally take Hemay007 tablets 600 mg BID for 12 weeks.
  Interventions: Drug: Hemay007
- placebo group (Placebo Comparator): Patients will orally take placebo tablets for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hemay007 — Hemay007 will be orally administered.
  Arms: Hemay007 400 mg BID group; Hemay007 600 mg BID group; Hemay007 800 mg QD group
Drug: Placebo — Placebo
  Arms: placebo group

SUMMARY:
This study adopts a multicenter, randomized, double-blind, low-medium-high dose group and placebo parallel controlled clinical study design. After screening, patients with active ulcerative colitis who meet the inclusion criteria and do not meet the exclusion criteria will be randomized by 1:1:1:1 to Hemay007 400 mg BID group, 800 mg QD group, 600 mg BID group or placebo group, with proposed 72 cases in each group. After 12 weeks of double-blind inductive treatment period, the patients will enter the Hemay007 open treatment period of 12 weeks when Hemay007 600 mg BID will be used as the medication regimen. All randomized subjects who have received the investigational drug should be subjected to a 4-week observation after the end of treatment.

DETAILED DESCRIPTION:
his study adopts a multicenter, randomized, double-blind, low-medium-high dose group and placebo parallel controlled clinical study design. After screening, patients with active ulcerative colitis who meet the inclusion criteria and do not meet the exclusion criteria will be randomized by 1:1:1:1 to Hemay007 400 mg BID group, 800 mg QD group, 600 mg BID group or placebo group, with proposed 72 cases in each group. After 12 weeks of double-blind inductive treatment period, the patients will enter the Hemay007 open treatment period of 12 weeks when Hemay007 600 mg BID will be used as the medication regimen. All randomized subjects who have received the investigational drug should be subjected to a 4-week observation after the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate in the trial and signing the informed consent forms;
* Age ≥18 years old and ≤70 years old, male or female;
* Diagnosed as ulcerative colitis (UC) ≥ 3 months at screening with clinical manifestations and evidence of endoscopy and confirmed by histopathological reports;
* Active ulcerative colitis with full Mayo score ≥ 4 points, and the subscore "endoscopic findings" in the Mayo endoscopic score within 14 days before randomization ≥ 2 points;
* UC treatment failure or intolerance (intolerance is defined as the discontinuation of drug use due to adverse reactions judged by the investigators) experienced by patients using at least one of the following:

Oral administration of sulfasalazine (SASP) and/or 5-aminosalicylic acid (5-ASA); Oral administration of corticosteroids; Azathioprine or 6-mercaptopurine; Anti-TNF-α treatment: infliximab or adalimumab, etc.;

* If the patient is using the following drugs to treat ulcerative colitis at the time of screening, it is necessary to receive stable treatment during the screening period and the following requirements during the study period are as follows:
* Oral administration of sulfasalazine (SASP) and/or 5-aminosalicylic acid (5-ASA) maintaining stable for at least ≥ 2 weeks prior to endoscopy during the screening period and maintaining stable during the study period; and/or
* Oral administration of low-dose corticosteroids (≤25 mg/d prednisolone or equivalent drug dose) maintaining stable for at least ≥ 2 weeks prior to endoscopy during the screening period;
* At least one of the following effective contraceptive methods should be adopted for female patients with fertility and male patients who have not undergone vasectomy during the entire study period from the date of signing the informed consent to 3 months after the last dose. Acceptable contraceptive methods in this study include: a. abstinence; b. hormones (oral intake, patch, ring, injection, implantation) combined with male condoms. This measure must be applied at least 30 days prior to the first administration of investigational drug, otherwise another acceptable method of contraception must be used; c. intra-uterine device (IUD) combined with male condoms; d. barrier method (diaphragm, cervical cap, sponge) combined with male condoms; exceptional circumstances: a) females who have been menopausal for 5 years and more, and b) surgical sterilization (proof should be provided).

Exclusion Criteria:

* Pregnant or lactating women, or women planning to become pregnant during the study;
* Knownto be allergic to any component of Hemay007 tablets (the main component is hemay007, and the main excipients are microcrystalline cellulose, pregelatinized starch, croscarmellose sodium, magnesium stearate);
* Patients with suspected or confirmed Crohn's disease, undiagnosed types of colitis, fulminant colitis, toxic megacolon, microscopic colitis, ischemic colitis or radioactive colitis based on medical history and endoscopy and/or histological results;
* Patients with the disease confined to the rectum (ulcerative proctitis) according to the endoscopy during screening;
* Patients who have undergone surgical treatment for ulcerative colitis or who require surgery during the study;
* Patientswith evidence of pathogenic intestinal infection;
* Patients receiving the following treatments:

Patients who have used azathioprine/6-mercaptopurine, methotrexate within 7 days before randomization; Patients who have used cyclosporine, mycophenolate mofetil, tacrolimus/sirolimus within 4 weeks before randomization; Patients who have used interferon within 8 weeks before randomization; Patients who have received anti-TNF-α treatment within 8 weeks before randomization; Intravenous corticosteroids or rectal administration of corticosteroids or rectal administration of 5-ASA within 2 weeks prior to randomization; Patients who have used thalidomide within 8 weeks before randomization;Patients who have received antibiotic treatment within 1 week before randomization;

• Patients with positive mycobacterium tuberculosis or potential mycobacterium tuberculosis infection, i.e. patients conforming to any one of the following definitions will be excluded: QuantiFERON®-TB Gold (QFT-G) or T-SPOT.TB test positive or purified protein derivative (PPD) skin test induration result ≥ 5 mm (within 3 months before screening); Chest imaging examination indicating positive tuberculosis (TB) infection lesion within 3 months prior to screening; History of latent or active TB infection;

* Patients with hemoglobin <8 g/dL or hematocrit <30%, white blood cells <3.0 × 10^9/L or neutrophils <1.2 × 10^9/L, platelets <100 × 10^09/L at screening;
* Total bilirubin (TBIL), aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥ 2 upper limits of normal (ULN) at screening;
* Glomerular filtration rate (eGFR) ≤ 40 ml/min;
* Patients with hereditary immunodeficiency disease;
* Patients with a history of lymphoproliferative disorders (e.g. EBV-related lymphoproliferative disorders), or with lymphoma, leukemia, myeloproliferative disease, multiple myeloma;
* Patients previously receiving drugs or treatment depleting lymphocytes (e.g. alemtuzumab, alkylating agents (e.g. cyclophosphamide or chlorambucil), total lymph node radiotherapy, etc.), however, patients can be enrolled if they used rituximab or other selective B lymphocyte depleting drugs more than one year before screening;
* Lymphocyte apheresis or selective mononuclear granulocyte apheresis was performed within 12 months before the screening or is planned to be performed during the study;
* The electrocardiogram during the screening period is abnormal and clinically significant, with the safety risk possibly increasing judged by the investigator;
* Blood donation ≥500 ml within 2 months before randomization;
* Patients with malignant tumor or with a history of malignancy other than well-treated or resected basal cell or squamous cell skin cancer;
* Patients with conditions that may affect oral drug absorption, e.g. gastrectomy or clinically significant diabetes-related gastrointestinal disorders, or specific types of obesity surgery such as gastric bypass, however, patients only subjected to the division of the stomach into independent chambers, like gastric banding, will not be excluded;
* Patients with previous surgery on small intestine or colon and with evidence of colonic dysplasia or intestinal stenosis; [21] Patients with chronic hepatitis B virus (HBV) infection (hepatitis B surface antigen (HBsAg), hepatitis B surface antibody (HBsAb) and hepatitis B core antibody (HBcAb) should be assessed for all patients during screening: patients with positive hepatitis B surface antigen (HBsAg) will be excluded; patients with HBsAg (negative), HBsAb (negative or positive) and HBcAb (positive) should be tested for HBV-DNA, and if the HBV-DNA result is positive, patient will be excluded; if the HBV-DNA result is negative, patients can be enrolled in the study.), chronic hepatitis C virus (HCV) infection (patients with positive hepatitis C virus antibody (HCVAb) excluded) or human immunodeficiency virus (HIV) infection (patients with positive human immunodeficiency virus (HIV) antibody excluded);
* Varicella, herpes zoster or other serious viral infections within 6 weeks prior to screening;
* Patients receive any live vaccine at present or has received any live vaccine within 8 weeks prior to randomization;
* Major organ transplantation (e.g. heart, lung, kidney, liver) or hematopoietic stem cell/bone marrow transplantation;
* Application of other drugs or devices of research nature within 3 months prior to randomization;
* Patients with primary sclerosing cholangitis;
* History of alcohol or drug abuse;
* Other conditions that the investigator judges as unsuitable to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-08-13 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2022-08-12 (Actual)

PRIMARY OUTCOMES:
clinical response | 12-week
  12-week clinical response rate Definition of clinical response: defined as full Mayo score decreased by ≥ 3 points compared with baseline and lowered by ≥ 30% compared with baseline, combined with the rectal bleeding subscore decreased by ≥ 1 point compared with baseline, or the absolute value of rectal bleeding subscore ≤ 1 point.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaowei Liu, M.D., Principal Investigator — XiangYa Hospital CentralSouth University
Locations (25):
- China (25):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Peking University International Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Army Special Medical Center, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Army Military Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Zhengzhou People's Hospital, Zhengzhou, Henan
  - Tongji hospital, tongji medical college, huazhong university of science and technology, Wuhan, Hubei
  - XiangYa Hospital CentralSouth University, Changsha, Hunan
  - Gulou Hospital Affiliated to Nanjing University School of Medicine, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Shengjing Hospital Affiliated to China Medical University, Shenyang, Liaoning
  - The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Neimenggu
  - Inner Mongolia Autonomous Region People's Hospital, Hohhot, Neimenggu
  - Affiliated Hospital of Qinghai University, Xining, Qinghai
  - Shandong Provincial Hospital, Jinan, Shandong
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
  - Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Shanxi Provincial People's Hospital, Taiyuan, Shanxi
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No